CLINICAL TRIAL: NCT06329297
Title: Continuous Glucose Monitoring in Medical and Open-Heart Surgical Patients
Brief Title: Continuous Glucose Monitoring in Inpatients
Status: Not yet recruiting | Type: Observational
Sponsor: Parkview Health (Other)
Responsible Party: Principal Investigator, Danielle Payne, FNP, Clinical Nurse Researcher & Nursing Research Program Coordinator, Parkview Health
Other Study IDs: NUR23-1005 INPTCGM1
Record Dates: First submitted 2024-03-01; First posted 2024-03-25 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hyperglycemia
Keywords: continuous glucose monitor; CGM
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Open-heart surgery inpatients: Patients having elective open-heart surgery including coronary artery bypass grafting (CABG), aortic valve repair/replacement (AVR), mitral valve repair/replacement (MVR), or any combination of those will have a CGM monitor placed within one hour of admission for up to 7 days or upon discharge.
  Interventions: Device: CGM monitor
- General medical inpatients: Medical inpatients who have a Glucommander order for management of hyperglycemia will have a CGM monitor placed within 24 hours of admission for up to 7 days or upon discharge.
  Interventions: Device: CGM monitor

INTERVENTIONS:
Device: CGM monitor — blood glucose sensor used to monitor interstitial glucose
  Other Names: Libre 3 Freestyle Continuous Glucose Monitor

SUMMARY:
The purpose of this study is to contribute to current research regarding the feasibility and accuracy of CGM in the hospital setting for both the medical and cardiovascular intensive care (ICU) patient populations.

DETAILED DESCRIPTION:
The use of continuous glucose monitors (CGM) in the outpatient setting has dramatically increased as these devices continue to improve in both ease of use, accessibility, and accuracy. Federal Drug Administration (FDA) clearance of certain devices has now been granted in both pregnancy and automated insulin delivery systems. As the world has embraced the safety and efficacy of continuous glucose monitors in the outpatient setting, health systems have turned attention to the potential of utilizing these devices to improve glycemic control in the hospital setting. With the announcement of the FDA granting enforcement discretion regarding the use of CGM technology in the hospital setting during the COVID-19 pandemic, the result was an abundance of research evaluating the potential of CGM longevity in the hospital setting.

The Standards of Care in Diabetes: 2023 reported that "preliminary data suggests that CGM can significantly improve glycemic management and other hospital outcomes." Additionally, a systematic review of 32 studies evaluated the accuracy of CGM in the intensive care unit, with a consensus of moderate to good accuracy. CGM in the hospital setting could provide a valuable tool in reducing hypoglycemia, hyperglycemia, and increasing time spent in normoglycemia. Other potential benefits of CGM include a broader view of glucose patterns, capture of asymptomatic hypoglycemia, reduced length of stay, and decreased cost. The Diabetes Technology Society organized the Hospital Consensus Guideline Panel in 2020, with the final report including the recommendation for additional research on the accuracy, data management, and patient-centered outcomes of CGM use in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients 18 years of age or older
* Glucose management per Glucommander and/or receiving POC blood glucose testing
* Patients admitted to Medical 6 or elective or urgent open-heart surgery patients admitted to the Cardiovascular Intensive Care Unit (CVICU)

Exclusion Criteria:

* Patients less than 18 years of age
* Pregnant or currently breastfeeding
* Prisoners
* Patients unable to consent in English.
* Patients with a preexisting insulin pump on admission
* Active skin infection at the insertion site(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients having elective open-heart surgery including coronary artery bypass grafting (CABG), aortic valve repair/replacement (AVR), mitral valve repair/replacement (MVR), or any combination of those and, Medical inpatients who have a Glucommander order for management of hyperglycemia.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CGM vs point of care test (POCT) glucose | from date of admission up to 7 days
  Continuous interstitial glucose monitor readings compared to point of care capillary blood glucose readings

SECONDARY OUTCOMES:
Slow downward trend arrow on CGM device | from date of admission up to 7 days
  impact on hypoglycemia events

CONTACTS AND LOCATIONS:
Overall Officials: Jan R Powers, Study Director — Parkview Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galindo RJ, Umpierrez GE, Rushakoff RJ, Basu A, Lohnes S, Nichols JH, Spanakis EK, Espinoza J, Palermo NE, Awadjie DG, Bak L, Buckingham B, Cook CB, Freckmann G, Heinemann L, Hovorka R, Mathioudakis N, Newman T, O'Neal DN, Rickert M, Sacks DB, Seley JJ, Wallia A, Shang T, Zhang JY, Han J, Klonoff DC. Continuous Glucose Monitors and Automated Insulin Dosing Systems in the Hospital Consensus Guideline. J Diabetes Sci Technol. 2020 Nov;14(6):1035-1064. doi: 10.1177/1932296820954163. Epub 2020 Sep 28. PMID 32985262
- [Background] van Steen SC, Rijkenberg S, Limpens J, van der Voort PH, Hermanides J, DeVries JH. The Clinical Benefits and Accuracy of Continuous Glucose Monitoring Systems in Critically Ill Patients-A Systematic Scoping Review. Sensors (Basel). 2017 Jan 14;17(1):146. doi: 10.3390/s17010146. PMID 28098809